CLINICAL TRIAL: NCT05071677
Title: Determinants of Treatment Decision Making in African American Women Diagnosed With Triple Negative Breast Cancer
Brief Title: Treatment Decision Making in African American Women Diagnosed With Triple Negative Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-1042; NCI-2021-09081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1042 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-23; First posted 2021-10-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Invasive Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey, interview): Patients participate in a standard of care treatment planning meeting over 3 hours with members of the multidisciplinary treatment team including, the oncologist, radiologist, oncology surgeon, and social worker. Patients then complete surveys over 20 minutes and within 30 days later. Some patients may participate in interviews over 30 minutes.
  Interventions: Procedure: Discussion; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Procedure: Discussion — Participate in treatment planning meeting
  Other Names: Discuss
Other: Interview — Participate in interview
Other: Survey Administration — Complete survey

SUMMARY:
This study evaluates what influences treatment decision-making in African American women with triple negative breast cancer. The study also aims to learn about the influence of information sources that support this decision-making process.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the acceptance of treatment recommendations by African American women diagnosed with triple negative breast cancer (TNBC).

SECONDARY OBJECTIVES:

I. Evaluate the association of beliefs about chemotherapy, self-efficacy, and cancer-specific psychological distress with intention to follow through with treatment.

II. Evaluate the association of intention, Reliance on Formal or Informal Resources, and decisional conflict as predictors of final treatment decision.

III. Evaluate the association of Reliance on Formal or Informal Resources as a moderator of the relationship between intention and final treatment decision.

OUTLINE:

Patients participate in a standard of care treatment planning meeting over 3 hours with members of the multidisciplinary treatment team including, the oncologist, radiologist, oncology surgeon, and social worker. Patients then complete surveys over 20 minutes and within 30 days later. Some patients may participate in interviews over 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* New patient in the MD Anderson Cancer Center Nellie B. Connally Breast Center or Houston Area Locations (HALs) (presenting to the surgery clinic, medical oncology clinic, or multiteam clinic)
* Women 18 years and older treated at MD Anderson Cancer Center between 1/1/2019 and 12/31/2021
* Diagnosis of triple negative invasive breast cancer on percutaneous needle biopsy within 60 days of first clinic appointment demonstrated by estrogen receptor (ER) 0% (absence or very low presence of estrogen uptake), progesterone receptor (PR) 0% (absence or very low presence of progesterone uptake), and HER2 negative (immunohistochemistry [IHC] score of 0 or 1 or fluorescence in situ hybridization [FISH] non-amplified score 2.0 or less)
* Tumor size >= 1 cm (chemotherapy is not recommended for tumors < 1 cm)
* Breast cancer stage I, II, or III
* Self-identify as of African descent (African American, African, Black, Afro-Caribbean, etc.)
* Completion of treatment planning team meeting and receipt of treatment at MD Anderson or local oncologist under the guidance of MD Anderson medical oncologist; no time window for treatment completion
* Ability to read, write, and speak in English, and provide consent

Exclusion Criteria:

* Patients with previous history of breast cancer diagnosis
* Patients with newly diagnosed bilateral breast cancer
* Patients with psychiatric disorders that exceed moderate severity documented within patient medical record

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of triple negative invasive breast
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who accept the recommended treatment plan | through study completion, an average of 1 year
  Patient demographics and clinical characteristics will be summarized using numerical summaries for continuous variables and proportions for categorical variables. The proportion of patients who accept the recommended treatment plan will be estimated along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Makesha V Miggins, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org